CLINICAL TRIAL: NCT01485328
Title: Phase III - Efficacy Study of AMARGOL - Phytomedicine on Therapeutics
Brief Title: Protocol: Phytomedicine-AMARGOL®, Clinical Trial for Efficacy Proof on Therapeutics
Acronym: AMARGOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorio Saude Ltda. (Industry)
Collaborators: Phytopharm Consulting Brazil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: labsaude-001-ama
Record Dates: First submitted 2008-12-16; First posted 2011-12-05 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Digestive System Disorders
Keywords: Dyspepsia; Flatulence; Aerophagia; Constipation
MeSH Terms: conditions — Digestive System Diseases; Dyspepsia; Flatulence; Aerophagy; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMARGOL (Active Comparator): per oral solution 40 mL single dose
  Interventions: Drug: AMARGOL®
- Vehicle without active principles (Placebo Comparator): per oral solution 40 mL single dose
  Interventions: Drug: AMARGOL®

INTERVENTIONS:
Drug: AMARGOL® — per oral solution, 40 mL single dose
  Other Names: AMARGOL; Phytomedicine; Herbal Extracts Mixture

SUMMARY:
This is a Phase 3: Efficacy Study for AMARGOL® a phytomedicine used for asymptomatic digestive complaints.

DETAILED DESCRIPTION:
This study will be performed for proving the efficacy of AMARGOL®, a phytomedicine product, under the Brazilian law for registration and revalidation RDC 14/2010.

AMARGOL® indications are for non specific digestive complaints as laxative and anti-dyspeptic.

Is a mixture of 7 plant extracts: Aloe ferox, Angelica archangelica, Alpinia officinarum, Cinnamomum zeylanicum, Gentiana lutea, Commiphora myrrh and Rheum palmatum.

Placebo controlled test

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* 65-85 Kg
* healthy volunteers

Exclusion Criteria:

* chronic dyspeptics illness chronic congestive cardiac problems
* pulmonary problems
* diabetes, thyroid problems
* pregnancy
* bowel syndrome
* hemorrhoids
* colitis
* allergies for any formula components.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
VAS - visual analogue scale | 24h
  Single dose 40mL AMARGOL 20 minutes before Dinner - strong meal

CONTACTS AND LOCATIONS:
Overall Officials: Angelo G Chaves, Doctor, Principal Investigator
Locations (1):
- Phytopharm Consulting, Porto Alegre, Rio Grande do Sul, Brazil